CLINICAL TRIAL: NCT01290172
Title: A Single-center, Randomized, Double Blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Somatostatin Used as Inflow Modulator in Liver Transplantation.
Brief Title: Evaluation of Efficacy and Safety of Somatostatin Used as Inflow Modulator in Liver Transplantation.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008/689; 2008-008319-24 (EudraCT Number)
Record Dates: First submitted 2011-02-03; First posted 2011-02-04 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Liver Transplant With Clinically Significant Portal Hypertension
Keywords: Liver transplant; portal hypertension
MeSH Terms: conditions — Hypertension, Portal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Somatostatin (Experimental): Patients in this group receive treatment with Somatostatin for 5 days.
  Interventions: Drug: Administration of Somatostatin
- Placebo (Placebo Comparator): Patients in this group receive a placebo for 5 days.
  Interventions: Drug: Administration of placebo

INTERVENTIONS:
Drug: Administration of Somatostatin — 6 mg will be diluted in saline in a 60 cc syringe to be infused over 24 h (250 mcg/h). The treatment will be started during the hepatectomy phase, after 1st measurement of native arterial and portal flow and pressure and given a clinically significant portal hypertension (CSPH) with a hepatic venous pressure gradient (HVPG) >= 10 mmHg.
  5 cc will be injected in 2 minutes as a single bolus of 500 mcg. Somatostatin will be given a second time at the beginning of the warm ischemia time as a continuous infusion of 250 mcg/h(infusion rate 2,5 cc/h). This will allow the time needed for reaching a stable plasma concentration at reperfusion and minimizing risks of secondary effects. After portal revascularization of the liver graft, a new measurement of portal flow and pressure will be performed. Provided a portal vein flow (PVF) >= 90 ml/min * 100 g LW, the remaining 55 cc will be infused for the following 22 h. 6 mg per day of continuous infusion will be continued for 5 days.
  Arms: Somatostatin
Drug: Administration of placebo — The placebo treatment will be started during the hepatectomy phase, after the 1st measurement of native arterial and portal flow and pressure and given a clinically significant portal hypertension (CSPH) with a hepatic venous pressure gradient (HVPG) >= 10 mmHg.
  5 cc of the 60 cc solution will be injected in 2 minutes as a single bolus of 500 mcg. The placebo will be given a 2nd time at the beginning of the warm ischemia time as a continuous infusion of 250 mcg/h (infusion rate 2,5 cc/h). This will allow the time needed for reaching a stable plasma concentration at reperfusion and minimizing risks of secondary effects. After portal revascularization of the liver graft, a new measurement of portal flow and pressure will be performed. Provided a portal vein flow (PVF) >= 90 ml/min * 100 gram LW, the remaining 55 cc will be infused for the following 22 h. 6 mg per day of continuous infusion will be continued everyday to complete 5 days of therapy.
  Arms: Placebo

SUMMARY:
This study is a 5 day, single-center, randomized, double blind, placebo-controlled study to evaluate the efficacy and safety of Somatostatin used as inflow modulator in liver transplantation. Patient systemic and hepatic dynamics will be collected and recorded at predefined time-points. To evaluate the ischemia-reperfusion injury, it is planned to perform liver biopsies at two different time-points to compare the liver structure and proteomic variations.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to provide written informed consent
* Cirrhotic patients with established clinically significant portal hypertension (CSPH) defined as an increase in hepatic venous pressure gradient >= 10 mmHg
* Recipients who are 18-70 years of age receiving a primary liver transplant from a brain dead donor or living donor
* Whole liver grafts and partial liver grafts can be included

Exclusion Criteria:

* Patients who are recipients of multiple solid organ transplants, or have previously received an organ or tissue transplant that may not be completely resolved by thrombectomy
* HIV positive patients
* Patients with known history of portal thrombosis or diagnosed at the time of transplantation that may not be completely resolved by thrombectomy.
* Patients included in the preoperative assessment without a CSPH at the time of the first intraoperative measurement of portal pressure
* Patients with low portal perfusion (=< 90 ml/min*100 g of LV) measured at the time of operation. Portal flows above this limit can be excluded in the eventuality that, after infusion, the portal perfusion falls below this limit
* Patients with porto-pulmonary hypertension
* Patients with known cardiac arrhythmias
* Recipients of cardiac-dead donors
* Fulminant hepatic failure patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2010-12; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of safety and efficacy using Somatostatin. | 5 days
  To evaluate the safety and efficacy, using Somatostatin as portal vein flow and pressure modulator in liver transplantation in humans. Hepatic and systemic hemodynamic measurements will be recorded prior, during and after the bolus infusion of Somatostatin/Placebo during liver transplantation. Infusion of Somatostatin/Placebo will be continued for 5 days.

SECONDARY OUTCOMES:
To elucidate pathophysiological pathways in non-cirrhotic grafted livers. | 35 days
To evaluate the reduction of ischemia-reperfusion injury (cytoprotective effect) | 1 hour after reperfusion and 5 days
To evaluate the efficacy of Somatostatin in the prevention of the small-for-size syndrome (SFSS) in partial liver transplantation. | after 35 days

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Troisi, PhD, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital, Ghent, Ghent, Belgium

REFERENCES:
- See also: Related Info — http://www.uzgent.be